CLINICAL TRIAL: NCT04258137
Title: Circulating DNA to Improve Outcome of Oncology PatiEnt: A Randomized Study - COPE Study
Brief Title: Circulating DNA to Improve Outcome of Oncology PatiEnt. A Randomized Study
Acronym: COPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IB 2019-06; 2019-A02479-48 (Other: ANSM IDRCB Number); ML41112 (Other: Roche ID)
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Colorectal Cancer; Non Small Cell Lung Cancer
Keywords: advanced; metastatic; liquid biopsy; genetic profiling
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — Liquid Biopsy

STUDY DESIGN:
Intervention Model Description: For each distinct population of patients with Advanced solid tumor (colorectal cancer and non-small-cell lung cancer), patients will be randomized between two arms:
  Experimental procedure: initial MTB providing therapeutic recommendation based on tumor sequencing and then follow-up combining standard imaging and ctDNA analysis (subsequent MTBs at each radiological assessment).
  Standard procedure: initial MTB providing therapeutic recommendation based on tumor sequencing and then follow-up based on standard imaging.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental procedure for colorectal cancer (Experimental): Patients with Advanced colorectal cancer will be managed by initial MTB providing therapeutic recommendation based on tumor sequencing and then follow-up combining standard imaging and ctDNA analysis (subsequent MTBs at each radiological assessment)
  Interventions: Genetic: Liquid biopsy
- Standard procedure for colorectal cancer (No Intervention): Patients with Advanced colorectal cancer will be managedby initial MTB providing therapeutic recommendation based on tumor sequencing and then follow-up based on standard imaging.
- Experimental procedure for non-small cell lung cancer (Experimental): Patients with Advanced non-small cell lung cancer will be managed by initial MTB providing therapeutic recommendation based on tumor sequencing and then follow-up combining standard imaging and ctDNA analysis (subsequent MTBs at each radiological assessment)
  Interventions: Genetic: Liquid biopsy
- Standard procedure for non-small cell lung cancer (No Intervention): Patients with Advanced non-small cell lung cancer will be managed by initial MTB providing therapeutic recommendation based on tumor sequencing and then follow-up based on standard imaging.

INTERVENTIONS:
Genetic: Liquid biopsy — Liquid biopsy will be performed at cycle 1 day 1 and cycle 2 day of each line of systemic treatment, at each tumor evaluation by Imaging and at confirmation of progression
  Arms: Experimental procedure for colorectal cancer; Experimental procedure for non-small cell lung cancer

SUMMARY:
COPE is a biology driven protocol with 2 independent, multicentric, two-arm non-comparative randomized (2:1) phase II trials in 2 distinct populations: colorectal cancer patients and non-small-lung cancer patients.

For each phase II trial, patient will be randomized between two arms with two patients randomized in arm A for one patient randomized in arm B:

* Arm A (Experimental - initial MTB providing therapeutic recommendation based on tumor sequencing and then follow-up combining standard imaging and ctDNA analysis)
* Arm B (Standard - initial MTB providing therapeutic recommendation based on tumor sequencing and then follow-up based on standard imaging).

DETAILED DESCRIPTION:
Primary tumor tissue, if accessible at all, does not always provide enough information to stratify individual patients to the most promising therapy. Re-analysis of metastatic lesions by needle biopsy is possible but invasive, and limited by the known intra-patient heterogeneity of individual lesions. These hurdles might be overcome by analyzing circulating tumor DNA (liquid biopsy), which in principle might reflect all subclones present at that specific time point and allow sequential monitoring of disease evolution.

Once tumor's genetic profiling is available, patients will be discussed within a multidisciplinary tumor board (MTB) which aims at discussing the genomic profiles and at providing a therapeutic decision for each patient. This MTB involves clinical oncologists, molecular biologists and clinical or biological project manager.

All the patients carrying an actionnable alteration will be proposed to receive a matched drug or to enter in a matched clinical trial depending on the possibility of inclusion at the time of molecular report.

the investigators hypothesize that implementing sequential circulating tumor DNA analysis can improve management of patients with advanced cancer and therefore their survival.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years,
2. Histology: colorectal cancer, non-small cell lung cancer,
3. Locally advanced/unresectable and/or metastatic solid tumor,
4. Eastern Cooperative Oncology Group (ECOG) performance status < 2 (Appendix 1),
5. Measurable disease according to RECIST 1.1 (lesion in previously irradiated filed can be considered as measurable if progressive at inclusion according to RECIST v1.1). At least one site of disease must be uni-dimensionally > 10 mm,
6. No previous systemic treatment for advanced disease,
7. Availability of suitable paraffin embedded (FFPE) archive tumor material or at least one target lesion that can be biopsied for research purpose,
8. Eligible to first-line systemic therapy,
9. Patient with a social security in compliance with the French law,
10. Voluntary signed and dated written informed consent prior to any study specific procedure.

Exclusion Criteria:

1. Inability to swallow,
2. Major problem with intestinal absorption,
3. Previous allogeneic bone marrow transplant,
4. Previous or current malignancies of other histologies within the last 2 years, with the exception of in situ carcinoma of the cervix, and adequately treated basal cell or squamous cell carcinoma of the skin and prostate cancer,
5. Evidence of severe or uncontrolled systemic disease (uncontrolled hypertension, active bleeding diatheses, or active Hepatitis B, C and HIV),
6. Any condition which in the Investigator's opinion makes it undesirable for the subject to participate in a clinical trial or which would jeopardize compliance with the protocol,
7. Individuals deprived of liberty or placed under guardianship,
8. Pregnant or breast feeding women,
9. Previous enrolment in the present study,
10. Any contraindication to first-line systemic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Estimated)
Dates: Start 2020-09-04 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of cancer outcome in terms of overall survival (2 distincts population) | 18 months
  Overall Survival (OS) is defined as the time interval between the date of randomization and the date of death (of any cause).

SECONDARY OUTCOMES:
Proportion of patients with at least one actionable alteration (in 2 distincts populations) | Throughout the study: an average of 18 months
  An actionable alteration is determined according to the molecular tumor board.
Proportion of patients treated with a targeted therapy (in 2 distincts populations) | Throughout the study: an average of 18 months
  A profiling-based targeted therapy corresponds to a therapy targeting an actionable alteration

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Centre hospitalier de la Côte Basque, Bayonne
  - Clinique Tivoli-Ducos, Bordeaux
  - Institut Bergonie, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - CHRU Brest, Brest
  - Polyclinique Marzet, Pau

IPD SHARING:
Plan to Share IPD: No